CLINICAL TRIAL: NCT03894540
Title: A Phase I, Open Label, Dose Escalation and Dose Expansion Study to Investigate the Safety, Pharmacokinetics, Pharmacodynamics and Anti-tumour Activity of IPN60090 as Single Agent and in Combination in Patients With Advanced Solid Tumours
Brief Title: Dose Escalation and Dose Expansion Study of IPN60090 in Patients With Advanced Solid Tumours
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Following an internal portfolio review, Ipsen has made the decision to terminate study D-US-60090-001. Ipsen would like to highlight that early termination was not due to any safety or tolerability issues with IPN60090
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D-US-60090-001; 2018-003681-13 (EudraCT Number)
Record Dates: First submitted 2019-03-27; First posted 2019-03-28 (Actual); Results first posted 2021-11-22 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-08

CONDITIONS: Solid Tumor
MeSH Terms: interventions — pembrolizumab; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- IPN60090 (Experimental): Part 1: Dose escalation of IPN60090, Part 2: Dose expansion
  IPN60090 given as a Bis in Die (BID) oral dose administered up to Maximum Tolerated Dose (MTD) over a 21-day cycle
  Interventions: Drug: IPN60090
- IPN60090 in combination with pembrolizumab (Experimental): Part 1: Dose escalation of IPN60090 in combination with pembrolizumab, Part 2: Dose expansion
  IPN60090 given as a Bis in Die (BID) oral dose, starting with pharmacologically active dose identified in 1dose escalation of IPN60090 as a single agent, over a 21-day cycle in combination with 200 mg pembrolizumab given every 21 days (Day 1 of every cycle) as IV infusion
  Interventions: Drug: IPN60090; Drug: pembrolizumab
- IPN60090 in combination with paclitaxel (Experimental): Part 1: Dose escalation of IPN60090 in combination with paclitaxel, Part 2: Dose expansion
  IPN60090 given as a BID oral dose, starting with pharmacologically active dose identified in dose escalation of IPN60090 as a single agent over a 21-day cycle in combination with 175 mg/m2 or 135 mg/m2 paclitaxel given every 21 days (Day 1 of every cycle) as IV infusion
  Interventions: Drug: IPN60090; Drug: paclitaxel
- IPN60090 food effect (Experimental): Part 1: Food Effect of IPN60090
  IPN60090 given as a single oral dose as a single agent at the recommended dose (RD) under fasting and fed conditions followed by IPN60090 given as a BID oral dose administered at the RD over a 21-day cycle.
  Interventions: Drug: IPN60090 single administration

INTERVENTIONS:
Drug: IPN60090 — Oral capsules given daily
  Arms: IPN60090; IPN60090 in combination with paclitaxel; IPN60090 in combination with pembrolizumab
Drug: pembrolizumab — An intravenous solution in single-use vial to be diluted for infusion.
  Arms: IPN60090 in combination with pembrolizumab
Drug: paclitaxel — An intravenous solution in single-use vial to be diluted for infusion.
  Arms: IPN60090 in combination with paclitaxel
Drug: IPN60090 single administration — Oral capsules given once
  Arms: IPN60090 food effect

SUMMARY:
The purpose of the protocol is to determine safety, tolerability, recommended dose (RD), pharmacokinetics (PK), pharmacodynamics (PD) and preliminary anti-tumour activity of IPN60090 as a single agent (Part A) and in combination with pembrolizumab (Part B) or paclitaxel (Part C) in patients with advanced solid tumours and to evaluate food effect (Part D).

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥18 years of age
* Patients with solid tumours who have received at least one line of therapy for advanced disease
* Measurable or non-measurable evaluable disease per RECIST 1.1
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) ≤1
* Standard of care and/or any investigational therapies must have been completed at least 3 weeks prior to treatment

Exclusion Criteria:

* Prior malignancy within the previous 2 years except for locally curable cancers that have been cured, such as basal or squamous cell skin cancer, or carcinoma in situ of the cervix, breast or bladder
* Known primary central malignancy or symptomatic central nervous system metastasis
* Major surgical intervention within 28 days before study drug administration
* Significant acute or chronic infections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-03-22 (Actual); Primary Completion 2020-12-21 (Actual); Study Completion 2020-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase 1 first in human dose escalation and dose expansion study was conducted in participants with advanced solid tumours at 1 investigational site in United States of America between 22 March 2019 and 21 December 2020. The sponsor decided to terminate the study during the dose escalation phase (Part A) of the study following an internal portfolio review.
Pre-assignment Details: The study was divided into 4 parts: Part A (dose escalation and dose expansion of IPN60090 monotherapy); Part B (dose escalation and dose expansion of IPN60090 + pembrolizumab); Part C (dose escalation and dose expansion of IPN60090 + paclitaxel); and Part D (food effect on IPN60090). Parts B, C and D were not performed due to study termination. A total of 22 participants received IPN60090 in Part A of the study.
Groups:
- IPN60090 20 mg: Participants received IPN60090 20 milligram (mg) capsules orally twice daily (BID) up to Cycle 7 in Part A of the study.
- IPN60090 40 mg: Participants received IPN60090 40 mg capsules orally BID up to Cycle 2 in Part A of the study.
- IPN60090 80 mg: Participants received IPN60090 80 mg capsules orally BID up to Cycle 5 in Part A of the study.
- IPN60090 120 mg: Participants received IPN60090 120 mg capsules orally BID up to Cycle 9 in Part A of the study.
- IPN60090 180 mg: Participants received IPN60090 180 mg capsules orally BID up to Cycle 9 in Part A of the study.
- IPN60090 240 mg: Participants received IPN60090 240 mg capsules orally BID up to Cycle 4 in Part A of the study.
Period: Overall Study
Arm/Group | IPN60090 20 mg | IPN60090 40 mg | IPN60090 80 mg | IPN60090 120 mg | IPN60090 180 mg | IPN60090 240 mg
Started (Received IPN60090 treatment in Part A.) | 1 | 1 | 1 | 4 | 11 | 4
Completed (Completed IPN60090 treatment in Part A.) | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 1 | 1 | 4 | 11 | 4
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Progressive Disease Per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 | 0 | 0 | 1 | 3 | 2 | 3
Not completed — Progressive Disease Clinical | 1 | 1 | 0 | 1 | 5 | 1
Not completed — Study termination by sponsor | 0 | 0 | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who were exposed to (or started receiving) IPN60090.
Groups:
- IPN60090 20 mg: Participants received IPN60090 20 mg capsules orally BID up to Cycle 7 in Part A of the study.
- Total: Total of all reporting groups
Arm/Group | IPN60090 20 mg | IPN60090 40 mg | IPN60090 80 mg | IPN60090 120 mg | IPN60090 180 mg | IPN60090 240 mg | Total
Number analyzed (Participants) | 1 | 1 | 1 | 4 | 11 | 4 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.0 (NA) — Standard deviation cannot be calculated when only one participant analyzed. | 47.0 (NA) — Standard deviation cannot be calculated when only one participant analyzed. | 63.0 (NA) — Standard deviation cannot be calculated when only one participant analyzed. | 57.0 (15.43) | 67.6 (7.15) | 47.8 (18.82) | 61.0 (13.49)
Age, Customized [Count of Participants; unit: Participants]
  16 to 64 years | 0 | 1 | 1 | 3 | 4 | 3 | 12
  65 to 84 years | 1 | 0 | 0 | 1 | 7 | 1 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1 | 4 | 6 | 4 | 16
  Male | 1 | 0 | 0 | 0 | 5 | 0 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Race: Black or African American | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Race: Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Race: White | 1 | 0 | 1 | 2 | 9 | 3 | 16
  Race: Other | 0 | 0 | 0 | 0 | 2 | 1 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 0 | 0 | 0 | 0 | 2 | 2 | 4
  Ethnicity: Not Hispanic or Latino | 1 | 1 | 1 | 4 | 9 | 2 | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (SAEs) in Part A
Description: An adverse event (AE) is the development of an undesirable medical condition or the deterioration of a pre-existing medical condition following or during exposure to a study drug, whether or not considered causally related to the study drug. An undesirable medical condition can be symptoms, signs or the abnormal results of an investigation. An SAE is any AE that: results in death; is life-threatening; requires hospitalization or prolongation of existing hospitalization; results in persistent or significant disability or incapacity; results in congenital anomaly or birth defect; or is medically important. A TEAE is defined as any AE that began or worsened following the first administration of study drugs. AEs were recorded and graded according of the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0.
  * Grade 1 = mild,
  * Grade 2 = moderate,
  * Grade 3 = severe,
  * Grade 4 = life threatening/disabling,
  * Grade 5 = death (related to AE).
Time Frame: TEAEs were to be collected from the start of the first dose of IPN60090 (Cycle 1 Day 1) up to 30 days after the date of the decision to permanently discontinue study treatment, assessed until data cut-off for study termination (maximum of 219 days).
Population: Safety population included all participants who were exposed to (or started receiving) IPN60090.
Measure: Count of Participants; unit: Participants
Arm/Group | IPN60090 20 mg | IPN60090 40 mg | IPN60090 80 mg | IPN60090 120 mg | IPN60090 180 mg | IPN60090 240 mg
Number analyzed (Participants) | 1 | 1 | 1 | 4 | 11 | 4
Participants
  Any TEAEs | 1 | 1 | 1 | 4 | 11 | 4
  TEAEs with NCI-CTCAE 5.0 Grade 3/4/5 | 1 | 1 | 1 | 2 | 8 | 3
  Treatment emergent SAEs | 1 | 0 | 1 | 2 | 4 | 3
  TEAEs leading to study treatment discontinuation | 0 | 0 | 0 | 0 | 1 | 0
  TEAEs leading to interruption or decrease of study treatment | 0 | 0 | 0 | 2 | 6 | 1
  TEAEs leading to interruption of study treatment | 0 | 0 | 0 | 2 | 6 | 1

2. Primary Outcome: Number of Participants With Dose-Limiting Toxicities (DLT) in Cycle 1 of Part A
Description: The maximum tolerated dose (MTD) is defined as the maximum dose of IPN60090 administered BID for 21 days, so that no more than 30% of participants experience a DLT. The MTD was determined using a Bayesian Optimal Interval design. The DLT assessment period was the first 21 days of treatment (one cycle).
Time Frame: Up to Cycle 1 Day 21 of Part A
Population: DLT evaluable population included all participants from the safety population who were evaluable for DLT (participants who completed at least one cycle of treatment and received ≥75% of the total planned dose of IPN60090 over the DLT assessment period).
Measure: Count of Participants; unit: Participants
Arm/Group | IPN60090 20 mg | IPN60090 40 mg | IPN60090 80 mg | IPN60090 120 mg | IPN60090 180 mg | IPN60090 240 mg
Number analyzed (Participants) | 1 | 1 | 1 | 4 | 11 | 4
Participants | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Recommended Dose of IPN60090 in Part A
Description: The recommended dose was determined by the safety review committee following an ad-hoc review of the safety and tolerability data during Part A of the study.
Time Frame: Up to Cycle 1 Day 21 of Part A
Population: as for outcome 2
Measure: Number; unit: mg
Groups:
- DLT Evaluable Population Analysis Set: DLT evaluable population included all participants from the safety population who were evaluable for DLT (participants who completed at least one cycle of treatment and received ≥75% of the total planned dose of IPN60090 over the DLT assessment period).
Arm/Group | DLT Evaluable Population Analysis Set
Number analyzed (Participants) | 22
mg | 180

4. Secondary Outcome: Best Overall Response (BOR) in Part A
Description: The BOR is defined as the best response designation [in the order of complete response (CR), partial response (PR), stable disease (SD), progressive disease (PD)] for each participant that is recorded between the date of the first dose of the study drug and the date of documented disease progression per RECIST 1.1 or the date of subsequent anticancer therapy whichever occurs first. Per RECIST v1.1, CR is disappearance of all target lesions; PR is >=30% decrease in the sum of the longest diameter of target lesions; and overall response = CR + PR.
Time Frame: RECIST assessments performed at baseline (within 28 days before start of study drug), every 6 weeks +/-1 week for first 24 weeks, then every 12 weeks +/-2 weeks thereafter. Up to data cut-off for study termination (maximum of 247 days).
Population: Efficacy population included all participants who received at least one dose of IPN60090.
Measure: Count of Participants; unit: Participants
Arm/Group | IPN60090 20 mg | IPN60090 40 mg | IPN60090 80 mg | IPN60090 120 mg | IPN60090 180 mg | IPN60090 240 mg
Number analyzed (Participants) | 1 | 1 | 1 | 4 | 11 | 4
Participants
  CR | 0 | 0 | 0 | 0 | 0 | 0
  PR | 0 | 0 | 0 | 0 | 0 | 0
  SD | 1 | 1 | 1 | 3 | 9 | 2
  PD | 0 | 0 | 0 | 1 | 2 | 2
  Not evaluable | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Objective Response Rate (ORR) in Part A
Description: The ORR is defined as the percentage of participants in whom the BOR is equal to CR and PR for Part A. The BOR is defined as the best response designation (in the order of CR, PR, SD, PD) for each participant that is recorded between the date of the first dose of the study drug and the date of documented disease progression per RECIST 1.1 or the date of subsequent anticancer therapy whichever occurs first. Per RECIST v1.1, CR is disappearance of all target lesions; PR is >=30% decrease in the sum of the longest diameter of target lesions; and overall response = CR + PR.
Time Frame: as for outcome 4
Population: Efficacy population included all participants who received at least one dose of IPN60090.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IPN60090 20 mg | IPN60090 40 mg | IPN60090 80 mg | IPN60090 120 mg | IPN60090 180 mg | IPN60090 240 mg
Number analyzed (Participants) | 1 | 1 | 1 | 4 | 11 | 4
percentage of participants | 0 [0.0 to 97.5] | 0 [0.0 to 97.5] | 0 [0.0 to 97.5] | 0 [0.0 to 60.2] | 0 [0.0 to 28.5] | 0 [0.0 to 60.2]

6. Secondary Outcome: Disease Control Rate (DCR) in Part A
Description: The DCR is defined as the percentage of participants in whom the BOR is equal to CR, PR or SD for Part A. The BOR is defined as the best response designation (in the order of CR, PR, SD, PD) for each participant that is recorded between the date of the first dose of the study drug and the date of documented disease progression per RECIST 1.1 or the date of subsequent anticancer therapy whichever occurs first. Per RECIST v1.1, CR is disappearance of all target lesions; PR is >=30% decrease in the sum of the longest diameter of target lesions; and overall response = CR + PR.
Time Frame: as for outcome 4
Population: Efficacy population included all participants who received at least one dose of IPN60090.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IPN60090 20 mg | IPN60090 40 mg | IPN60090 80 mg | IPN60090 120 mg | IPN60090 180 mg | IPN60090 240 mg
Number analyzed (Participants) | 1 | 1 | 1 | 4 | 11 | 4
percentage of participants | 100.0 [2.5 to 100.0] | 100.0 [2.5 to 100.0] | 100.0 [2.5 to 100.0] | 75.0 [19.4 to 99.4] | 81.8 [48.2 to 97.7] | 50.0 [6.8 to 93.2]

7. Secondary Outcome: Mean Progression Free Survival (PFS) in Part A
Description: The PFS is defined as the time from first dose of study drug to the first documented objective disease progression (for RECIST 1.1), clinical disease progression collected at end of treatment, or death due to any cause, whichever occurred first. Per RECIST 1.1, progression is defined as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: as for outcome 4
Population: Efficacy population included all participants who received at least one dose of IPN60090.
Measure: Mean (Standard Deviation); unit: months
Arm/Group | IPN60090 20 mg | IPN60090 40 mg | IPN60090 80 mg | IPN60090 120 mg | IPN60090 180 mg | IPN60090 240 mg
Number analyzed (Participants) | 1 | 1 | 1 | 4 | 11 | 4
months | 4.90 (NA) — Standard deviation cannot be calculated when only one participant analyzed. | 1.45 (NA) — Standard deviation cannot be calculated when only one participant analyzed. | 2.73 (NA) — Standard deviation cannot be calculated when only one participant analyzed. | 2.81 (2.193) | 4.37 (2.766) | 1.52 (0.073)

8. Secondary Outcome: Mean Overall Survival (OS) in Part A
Description: The OS is defined as the time from first dose of study drug to death due to any cause. Participants who were lost to follow-up or who were still alive at the time of analysis is censored at the last day the participant was known to be alive or data cut-off date, whichever occurred first.
Time Frame: as for outcome 4
Population: Efficacy population included all participants who received at least one dose of IPN60090.
Measure: Mean (Standard Deviation); unit: months
Arm/Group | IPN60090 20 mg | IPN60090 40 mg | IPN60090 80 mg | IPN60090 120 mg | IPN60090 180 mg | IPN60090 240 mg
Number analyzed (Participants) | 1 | 1 | 1 | 4 | 11 | 4
months | 5.03 (NA) — Standard deviation cannot be calculated when only one participant analyzed. | 6.21 (NA) — Standard deviation cannot be calculated when only one participant analyzed. | 13.24 (NA) — Standard deviation cannot be calculated when only one participant analyzed. | 6.35 (4.433) | 11.00 (5.421) | 11.01 (4.409)

9. Secondary Outcome: Mean Best Percent Change From Baseline in the Sum of Diameters of the Target Lesions at Minimum Post-Baseline in Part A
Description: All measurable lesions up to a maximum of two lesions per organ and five lesions in total, representative of all involved organs, identified as target lesions and measured at baseline. Baseline is defined as the last measurement prior to the first dose of study drug.
Time Frame: Baseline (within 28 days before start of study drug) and post-baseline, up to data cut-off for study termination (maximum of 247 days).
Population: Efficacy population included all participants who received at least one dose of IPN60090. Only participants with valid baseline and at least one post-baseline value of the sum of diameters are included.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | IPN60090 20 mg | IPN60090 40 mg | IPN60090 80 mg | IPN60090 120 mg | IPN60090 180 mg | IPN60090 240 mg
Number analyzed (Participants) | 1 | 1 | 1 | 2 | 9 | 4
percent change | 0.0 (NA) — Standard deviation cannot be calculated when only one participant analyzed. | 7.7 (NA) — Standard deviation cannot be calculated when only one participant analyzed. | -21.6 (NA) — Standard deviation cannot be calculated when only one participant analyzed. | -10.2 (14.48) | 3.6 (18.05) | 18.3 (20.88)

10. Secondary Outcome: Maximum Observed Concentration (Cmax) of IPN60090 in Part A
Description: Blood samples were collected to determine Cmax of IPN60090. The pharmacokinetics (PK) of IPN60090 plasma concentrations were performed using noncompartmental analysis.
Time Frame: Pre-dose and 0.5, 1, 2, 4, 8 and 12 hours post-dose on Cycle 1 Day 1 and Cycle 1 Day 14 in Part A
Population: The PK population for noncompartmental analysis included all participants who had no major protocol deviation affecting the PK variables and who had a sufficient number of IPN60090 plasma concentrations to estimate the main PK parameters. Summarized PK results are presented for IPN60090 120 mg, IPN60090 180 mg and IPN60090 240 mg reporting groups only.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | IPN60090 120 mg | IPN60090 180 mg | IPN60090 240 mg
Number analyzed (Participants) | 4 | 11 | 4
nanogram per milliliter (ng/mL)
  Cycle 1 Day 1 | 10019 (4429) | 13467 (8780) | 13068 (11503)
  Cycle 1 Day 14: number analyzed (Participants) | 3 | 9 | 4
  Cycle 1 Day 14 | 19595 (16103) | 24395 (9912) | 25793 (16215)

11. Secondary Outcome: Time to Reach Maximum Observed Concentration (Tmax) of IPN60090 in Part A
Description: Blood samples were collected to determine Tmax of IPN60090. The PK of IPN60090 plasma concentrations were performed using noncompartmental analysis.
Time Frame: Pre-dose and 0.5, 1, 2, 4, 8 and 12 hours post-dose on Cycle 1 Day 1 and Cycle 1 Day 14 in Part A
Population: as for outcome 10
Measure: Median (Full Range); unit: hours
Arm/Group | IPN60090 120 mg | IPN60090 180 mg | IPN60090 240 mg
Number analyzed (Participants) | 4 | 11 | 4
hours
  Cycle 1 Day 1 | 2.10 [1.00 to 4.08] | 4.00 [1.00 to 4.17] | 4.04 [1.08 to 4.13]
  Cycle 1 Day 14: number analyzed (Participants) | 3 | 9 | 4
  Cycle 1 Day 14 | 1.00 [0.93 to 2.00] | 2.00 [1.00 to 4.08] | 1.58 [0.00 to 4.00]

12. Secondary Outcome: Trough Plasma Concentration (Ctrough) of IPN60090 in Part A
Description: Blood samples were collected to determine Ctrough of IPN60090. The PK of IPN60090 plasma concentrations were performed using noncompartmental analysis.
Time Frame: Pre-dose and 0.5, 1, 2, 4, 8 and 12 hours post-dose on Cycle 1 Day 14 in Part A
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | IPN60090 120 mg | IPN60090 180 mg | IPN60090 240 mg
Number analyzed (Participants) | 3 | 9 | 4
ng/mL | 9211 (8149) | 14616 (6654) | 20214 (15970)

13. Secondary Outcome: Area Under the Concentration Versus Time Curve From Time Zero to the Last Quantifiable Concentration (AUC0-last) of IPN60090 in Part A
Description: Blood samples were collected to determine AUC0-last of IPN60090. The PK of IPN60090 plasma concentrations were performed using noncompartmental analysis.
Time Frame: Pre-dose and 0.5, 1, 2, 4, 8 and 12 hours post-dose on Cycle 1 Day 1 and Cycle 1 Day 14 in Part A
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: hour*ng/mL
Arm/Group | IPN60090 120 mg | IPN60090 180 mg | IPN60090 240 mg
Number analyzed (Participants) | 4 | 11 | 4
hour*ng/mL
  Cycle 1 Day 1 | 62776 (31857) | 87061 (54015) | 67192 (54492)
  Cycle 1 Day 14: number analyzed (Participants) | 3 | 9 | 4
  Cycle 1 Day 14 | 128699 (99755) | 188838 (91394) | 200845 (128710)

14. Secondary Outcome: Apparent Elimination Half-Life (T1/2) of IPN60090 in Part A
Description: Blood samples were collected to determine T1/2 of IPN60090. The PK of IPN60090 plasma concentrations were performed using noncompartmental analysis.
Time Frame: Pre-dose and 0.5, 1, 2, 4, 8 and 12 hours post-dose on Cycle 1 Day 1 in Part A
Population: as for outcome 10
Measure: Median (Full Range); unit: hours
Arm/Group | IPN60090 120 mg | IPN60090 180 mg | IPN60090 240 mg
Number analyzed (Participants) | 3 | 4 | 1
hours | 12.72 [9.01 to 25.48] | 6.92 [5.85 to 10.87] | 6.18 [6.18 to 6.18]

15. Secondary Outcome: Apparent Total Body Clearance (CL/F) of IPN60090 in Part A
Description: Blood samples were collected to determine CL/F of IPN60090. The PK of IPN60090 plasma concentrations were performed using noncompartmental analysis.
Time Frame: Pre-dose and 0.5, 1, 2, 4, 8 and 12 hours post-dose on Cycle 1 Day 1 in Part A
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: liter per hour
Arm/Group | IPN60090 120 mg | IPN60090 180 mg | IPN60090 240 mg
Number analyzed (Participants) | 3 | 4 | 1
liter per hour | 0.811 (0.190) | 1.03 (0.270) | 3.71 (NA) — Standard deviation cannot be calculated when only one participant analyzed.

16. Secondary Outcome: Apparent Volume of Distribution (Vz/F) of IPN60090 in Part A
Description: Blood samples were collected to determine Vz/F of IPN60090. The PK of IPN60090 plasma concentrations were performed using noncompartmental analysis.
Time Frame: Pre-dose and 0.5, 1, 2, 4, 8 and 12 hours post-dose on Cycle 1 Day 1 in Part A
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: liter
Arm/Group | IPN60090 120 mg | IPN60090 180 mg | IPN60090 240 mg
Number analyzed (Participants) | 3 | 4 | 1
liter | 20.0 (15.5) | 11.2 (3.35) | 33.0 (NA) — Standard deviation cannot be calculated when only one participant analyzed.

17. Secondary Outcome: Target Engagement in Part A
Description: The target engagement is glutamate:glutamine (Glu:Gln) ratio in peripheral blood mononuclear cells. Glu:Gln ratio inhibition is calculated as (1 - post-baseline Glu:Gln ratio/Cycle 1 Day 1 predose Glu:Gln ratio) x 100%.
Time Frame: At 2 and 12 hours postdose on Cycle 1 Day 1; predose, 2 and 12 hours postdose on Cycle 1 Day 14; and predose, 2 and 2-4 hours postdose on Cycle 1 Day 15 in Part A
Population: Efficacy population included all participants who received at least one dose of IPN60090.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | IPN60090 20 mg | IPN60090 40 mg | IPN60090 80 mg | IPN60090 120 mg | IPN60090 180 mg | IPN60090 240 mg
Number analyzed (Participants) | 1 | 1 | 1 | 4 | 11 | 4
ratio
  Cycle 1 Day 1: 2 hours postdose: number analyzed (Participants) | 0 | 1 | 1 | 3 | 7 | 4
  Cycle 1 Day 1: 2 hours postdose |  | 75.66 (NA) — Standard deviation cannot be calculated when only one participant analyzed. | 67.06 (NA) — Standard deviation cannot be calculated when only one participant analyzed. | 85.02 (8.734) | 86.13 (7.216) | 82.65 (14.286)
  Cycle 1 Day 1: 12 hours postdose: number analyzed (Participants) | 0 | 1 | 1 | 3 | 7 | 4
  Cycle 1 Day 1: 12 hours postdose |  | 61.90 (NA) — Standard deviation cannot be calculated when only one participant analyzed. | 34.12 (NA) — Standard deviation cannot be calculated when only one participant analyzed. | 72.47 (19.188) | 75.43 (17.521) | 70.94 (18.055)
  Cycle 1 Day 14: predose: number analyzed (Participants) | 1 | 1 | 1 | 2 | 6 | 4
  Cycle 1 Day 14: predose | 50.45 (NA) — Standard deviation cannot be calculated when only one participant analyzed. | 36.51 (NA) — Standard deviation cannot be calculated when only one participant analyzed. | 80.42 (NA) — Standard deviation cannot be calculated when only one participant analyzed. | 82.59 (12.622) | 83.15 (11.554) | 83.12 (10.962)
  Cycle 1 Day 14: 2 hours postdose: number analyzed (Participants) | 1 | 1 | 1 | 2 | 5 | 4
  Cycle 1 Day 14: 2 hours postdose | 65.77 (NA) — Standard deviation cannot be calculated when only one participant analyzed. | 75.66 (NA) — Standard deviation cannot be calculated when only one participant analyzed. | 84.42 (NA) — Standard deviation cannot be calculated when only one participant analyzed. | 88.30 (7.798) | 91.83 (3.099) | 87.48 (6.257)
  Cycle 1 Day 14: 12 hours postdose: number analyzed (Participants) | 1 | 1 | 1 | 2 | 5 | 4
  Cycle 1 Day 14: 12 hours postdose | 50.45 (NA) — Standard deviation cannot be calculated when only one participant analyzed. | 69.31 (NA) — Standard deviation cannot be calculated when only one participant analyzed. | 84.87 (NA) — Standard deviation cannot be calculated when only one participant analyzed. | 82.00 (13.609) | 86.51 (5.474) | 74.38 (22.991)
  Cycle 1 Day 15: predose: number analyzed (Participants) | 1 | 1 | 1 | 2 | 5 | 4
  Cycle 1 Day 15: predose | 72.07 (NA) — Standard deviation cannot be calculated when only one participant analyzed. | 56.61 (NA) — Standard deviation cannot be calculated when only one participant analyzed. | 72.40 (NA) — Standard deviation cannot be calculated when only one participant analyzed. | 87.25 (4.898) | 86.67 (3.767) | 86.67 (9.394)
  Cycle 1 Day 15: 2 hours postdose: number analyzed (Participants) | 1 | 1 | 1 | 0 | 2 | 0
  Cycle 1 Day 15: 2 hours postdose | 79.28 (NA) — Standard deviation cannot be calculated when only one participant analyzed. | 71.43 (NA) — Standard deviation cannot be calculated when only one participant analyzed. | 79.97 (NA) — Standard deviation cannot be calculated when only one participant analyzed. |  | 89.57 (3.125) |
  Cycle 1 Day 15: 2-4 hours postdose: number analyzed (Participants) | 0 | 0 | 0 | 2 | 2 | 4
  Cycle 1 Day 15: 2-4 hours postdose |  |  |  | 88.35 (5.721) | 88.73 (4.517) | 88.16 (6.123)

ADVERSE EVENTS:
Time Frame: TEAEs were to be collected from the start of the first dose of IPN60090 (Cycle 1 Day 1) up to 30 days after the date of the decision to permanently discontinue study treatment, assessed until data cut-off for study termination (maximum of 219 days).
Description: Safety population included all participants who were exposed to (or started receiving) IPN60090.
Arm/Group | IPN60090 20 mg | IPN60090 40 mg | IPN60090 80 mg | IPN60090 120 mg | IPN60090 180 mg | IPN60090 240 mg
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1 | 0/1 | 0/4 | 0/11 | 0/4
Serious Adverse Events (participants affected / at risk) | 1/1 | 0/1 | 1/1 | 2/4 | 4/11 | 3/4
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 1/1 | 4/4 | 11/11 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IPN60090 20 mg (N=1) | IPN60090 40 mg (N=1) | IPN60090 80 mg (N=1) | IPN60090 120 mg (N=4) | IPN60090 180 mg (N=11) | IPN60090 240 mg (N=4)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aeromonas infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cryptosporidiosis infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Brain oedema (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Biliary obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IPN60090 20 mg (N=1) | IPN60090 40 mg (N=1) | IPN60090 80 mg (N=1) | IPN60090 120 mg (N=4) | IPN60090 180 mg (N=11) | IPN60090 240 mg (N=4)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 3 (3) | 3 (7)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (3)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (6) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oesophageal stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (11) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 1 (4) | 1 (4)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Photopsia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (6) | 1 (1)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 2 (2)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vitreous floaters (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Migraine with aura (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Facial paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (3)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (3)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 4 (9) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 2 (6)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (6) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (7) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 2 (3)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was terminated by the sponsor following an internal portfolio review during the dose escalation phase (Part A). The early termination was not due to any safety or tolerability issues with IPN60090.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-12-10): https://cdn.clinicaltrials.gov/large-docs/40/NCT03894540/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-17): https://cdn.clinicaltrials.gov/large-docs/40/NCT03894540/SAP_001.pdf